CLINICAL TRIAL: NCT06084195
Title: Unravelling Tumour Biology In Ovarian Cancer With Precision Imaging
Acronym: MR-O-MICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2023-02 MRO
Record Dates: First submitted 2023-10-02; First posted 2023-10-16 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: High Grade Serous Ovarian Cancer
Keywords: Radiomics; Ovarian cancer; Genomics; Proteomics; Immune Tumor Microenvironment
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Blood Specimen Collection; Histocompatibility Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): single arm
  Interventions: Biological: Blood sample and tissue sample

INTERVENTIONS:
Biological: Blood sample and tissue sample — During the surgery :
  * Tissus sample : primary tumor and metastasis
  * blood sample : 3 EDTA tubes
  * ex vivo MRI data

SUMMARY:
The objective of this study is to explore the integration of in vivo and ex vivo of MRI with histology and molecular assessments to advance non-invasive characterization of tumor heterogeneity in high-grade serous ovarian cance

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patient giving wirtting informed consent.

During surgery, tissue and blood samples will be conserved for the study. In this study will be compared images obtained in vivo before surgical management, ex vivo images obtained on excised tissues during surgery, histological data obtained during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged >18
* Pathologically proven HGSOC at an advanced stage (FIGO IIIB or IIIC) which can benefit from surgery with or without prior neoadjuvant treatment
* Willingness and ability to comply with planned visits, treatment plan, laboratory tests and other study procedures,
* Patient who has given informed, written and express consent,
* Patient affiliated with a French health insurance scheme.

Exclusion Criteria:

* Early-stage disease (FIGO <IIIB) or presence of extraperitoneal metastases,
* Patient who will not have surgery
* Patient whose regular follow-up is impossible for psychological, family, social or geographical reasons,
* Patient under guardianship, curatorship or safeguarding of justice,
* Pregnant and/or nursing patient,
* Patient with a history of other cancers within 5 years/10 years prior to inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
the integration of in vivo and ex vivo of MRI with histology and molecular assessments to advance non-invasive characterization of tumor heterogeneity in high-grade serous ovarian cancer. | one shoot at the surgery
  The diagnostic performance of the radiomic and multiomic algorithm for the characterization of heterogeneity in the CSOHG.

SECONDARY OUTCOMES:
the imaging phenotype of tumor heterogeneity with a multi-scale radiomic approach by obtaining the image mirror tumor at the in vivo scale | one shoot at the surgery
  Correlation between radiomic maps and pathogenic maps of heterogeneity,
tumor heterogeneity based on phenotypic imaging supported by AI reflects and can predict sub-histologyunderlying by tumor stroma proportion and tumor density infiltrating lymphocytes and genomics through HRD | one shoot at the surgery
  Correlation between radiomic algorithms and i/underlying histology and ii/ genomics
the heterogeneity of the tumor biology of CSOHG through non-invasive habitat imaging combined with an integrated Multi-O-Mics approach. | one shoot at the surgery
  Correlation between radiomic maps and tumor biology (CYTOF, proteomics and transcriptomics),
To Correlate MRI results with hematological molecular biology results. | one shoot at the surgery
  Correlation between radiomic algorithms for tumor detection and cDNA determination.

CONTACTS AND LOCATIONS:
Overall Officials: NOUGARET Stephanie, MD, Study Director — INSTITUT REGIONAL DU CANCER DE MONTPELLIER Cancer de Montpellier
Locations (1):
- NOUGARET Stephanie, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torre LA, Trabert B, DeSantis CE, Miller KD, Samimi G, Runowicz CD, Gaudet MM, Jemal A, Siegel RL. Ovarian cancer statistics, 2018. CA Cancer J Clin. 2018 Jul;68(4):284-296. doi: 10.3322/caac.21456. Epub 2018 May 29. PMID 29809280
- [Background] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Background] Vergote I, Trope CG, Amant F, Kristensen GB, Ehlen T, Johnson N, Verheijen RH, van der Burg ME, Lacave AJ, Panici PB, Kenter GG, Casado A, Mendiola C, Coens C, Verleye L, Stuart GC, Pecorelli S, Reed NS; European Organization for Research and Treatment of Cancer-Gynaecological Cancer Group; NCIC Clinical Trials Group. Neoadjuvant chemotherapy or primary surgery in stage IIIC or IV ovarian cancer. N Engl J Med. 2010 Sep 2;363(10):943-53. doi: 10.1056/NEJMoa0908806. PMID 20818904
- [Background] van Driel WJ, Koole SN, Sikorska K, Schagen van Leeuwen JH, Schreuder HWR, Hermans RHM, de Hingh IHJT, van der Velden J, Arts HJ, Massuger LFAG, Aalbers AGJ, Verwaal VJ, Kieffer JM, Van de Vijver KK, van Tinteren H, Aaronson NK, Sonke GS. Hyperthermic Intraperitoneal Chemotherapy in Ovarian Cancer. N Engl J Med. 2018 Jan 18;378(3):230-240. doi: 10.1056/NEJMoa1708618. PMID 29342393
- [Background] Jayson GC, Kohn EC, Kitchener HC, Ledermann JA. Ovarian cancer. Lancet. 2014 Oct 11;384(9951):1376-88. doi: 10.1016/S0140-6736(13)62146-7. Epub 2014 Apr 21. PMID 24767708
- [Background] Cancer Genome Atlas Research Network. Integrated genomic analyses of ovarian carcinoma. Nature. 2011 Jun 29;474(7353):609-15. doi: 10.1038/nature10166. PMID 21720365
- [Background] Cooke SL, Brenton JD. Evolution of platinum resistance in high-grade serous ovarian cancer. Lancet Oncol. 2011 Nov;12(12):1169-74. doi: 10.1016/S1470-2045(11)70123-1. PMID 21742554
- [Background] McPherson A, Roth A, Laks E, Masud T, Bashashati A, Zhang AW, Ha G, Biele J, Yap D, Wan A, Prentice LM, Khattra J, Smith MA, Nielsen CB, Mullaly SC, Kalloger S, Karnezis A, Shumansky K, Siu C, Rosner J, Chan HL, Ho J, Melnyk N, Senz J, Yang W, Moore R, Mungall AJ, Marra MA, Bouchard-Cote A, Gilks CB, Huntsman DG, McAlpine JN, Aparicio S, Shah SP. Divergent modes of clonal spread and intraperitoneal mixing in high-grade serous ovarian cancer. Nat Genet. 2016 Jul;48(7):758-67. doi: 10.1038/ng.3573. Epub 2016 May 16. PMID 27182968
- [Background] Burrell RA, Swanton C. Tumour heterogeneity and the evolution of polyclonal drug resistance. Mol Oncol. 2014 Sep 12;8(6):1095-111. doi: 10.1016/j.molonc.2014.06.005. Epub 2014 Jul 10. PMID 25087573
- [Background] Hoogstraat M, de Pagter MS, Cirkel GA, van Roosmalen MJ, Harkins TT, Duran K, Kreeftmeijer J, Renkens I, Witteveen PO, Lee CC, Nijman IJ, Guy T, van 't Slot R, Jonges TN, Lolkema MP, Koudijs MJ, Zweemer RP, Voest EE, Cuppen E, Kloosterman WP. Genomic and transcriptomic plasticity in treatment-naive ovarian cancer. Genome Res. 2014 Feb;24(2):200-11. doi: 10.1101/gr.161026.113. Epub 2013 Nov 12. PMID 24221193
- [Background] Lee JY, Yoon JK, Kim B, Kim S, Kim MA, Lim H, Bang D, Song YS. Tumor evolution and intratumor heterogeneity of an epithelial ovarian cancer investigated using next-generation sequencing. BMC Cancer. 2015 Feb 26;15:85. doi: 10.1186/s12885-015-1077-4. PMID 25881093
- [Background] Schwarz RF, Ng CK, Cooke SL, Newman S, Temple J, Piskorz AM, Gale D, Sayal K, Murtaza M, Baldwin PJ, Rosenfeld N, Earl HM, Sala E, Jimenez-Linan M, Parkinson CA, Markowetz F, Brenton JD. Spatial and temporal heterogeneity in high-grade serous ovarian cancer: a phylogenetic analysis. PLoS Med. 2015 Feb 24;12(2):e1001789. doi: 10.1371/journal.pmed.1001789. eCollection 2015 Feb. PMID 25710373
- [Background] Bashashati A, Ha G, Tone A, Ding J, Prentice LM, Roth A, Rosner J, Shumansky K, Kalloger S, Senz J, Yang W, McConechy M, Melnyk N, Anglesio M, Luk MT, Tse K, Zeng T, Moore R, Zhao Y, Marra MA, Gilks B, Yip S, Huntsman DG, McAlpine JN, Shah SP. Distinct evolutionary trajectories of primary high-grade serous ovarian cancers revealed through spatial mutational profiling. J Pathol. 2013 Sep;231(1):21-34. doi: 10.1002/path.4230. PMID 23780408
- [Background] Greaves M, Maley CC. Clonal evolution in cancer. Nature. 2012 Jan 18;481(7381):306-13. doi: 10.1038/nature10762. PMID 22258609
- [Background] Zhang AW, McPherson A, Milne K, Kroeger DR, Hamilton PT, Miranda A, Funnell T, Little N, de Souza CPE, Laan S, LeDoux S, Cochrane DR, Lim JLP, Yang W, Roth A, Smith MA, Ho J, Tse K, Zeng T, Shlafman I, Mayo MR, Moore R, Failmezger H, Heindl A, Wang YK, Bashashati A, Grewal DS, Brown SD, Lai D, Wan ANC, Nielsen CB, Huebner C, Tessier-Cloutier B, Anglesio MS, Bouchard-Cote A, Yuan Y, Wasserman WW, Gilks CB, Karnezis AN, Aparicio S, McAlpine JN, Huntsman DG, Holt RA, Nelson BH, Shah SP. Interfaces of Malignant and Immunologic Clonal Dynamics in Ovarian Cancer. Cell. 2018 Jun 14;173(7):1755-1769.e22. doi: 10.1016/j.cell.2018.03.073. Epub 2018 May 10. PMID 29754820
- [Background] Jimenez-Sanchez A, Memon D, Pourpe S, Veeraraghavan H, Li Y, Vargas HA, Gill MB, Park KJ, Zivanovic O, Konner J, Ricca J, Zamarin D, Walther T, Aghajanian C, Wolchok JD, Sala E, Merghoub T, Snyder A, Miller ML. Heterogeneous Tumor-Immune Microenvironments among Differentially Growing Metastases in an Ovarian Cancer Patient. Cell. 2017 Aug 24;170(5):927-938.e20. doi: 10.1016/j.cell.2017.07.025. PMID 28841418
- [Background] Jimenez-Sanchez A, Cybulska P, Mager KL, Koplev S, Cast O, Couturier DL, Memon D, Selenica P, Nikolovski I, Mazaheri Y, Bykov Y, Geyer FC, Macintyre G, Gavarro LM, Drews RM, Gill MB, Papanastasiou AD, Sosa RE, Soslow RA, Walther T, Shen R, Chi DS, Park KJ, Hollmann T, Reis-Filho JS, Markowetz F, Beltrao P, Vargas HA, Zamarin D, Brenton JD, Snyder A, Weigelt B, Sala E, Miller ML. Unraveling tumor-immune heterogeneity in advanced ovarian cancer uncovers immunogenic effect of chemotherapy. Nat Genet. 2020 Jun;52(6):582-593. doi: 10.1038/s41588-020-0630-5. Epub 2020 Jun 1. PMID 32483290
- [Background] Frey MK, Pothuri B. Homologous recombination deficiency (HRD) testing in ovarian cancer clinical practice: a review of the literature. Gynecol Oncol Res Pract. 2017 Feb 22;4:4. doi: 10.1186/s40661-017-0039-8. eCollection 2017. PMID 28250960
- [Background] Yildirim N, Akman L, Acar K, Demir S, Ozkan S, Alan N, Zekioglu O, Terek MC, Ozdemir N, Ozsaran A. Do tumor-infiltrating lymphocytes really indicate favorable prognosis in epithelial ovarian cancer? Eur J Obstet Gynecol Reprod Biol. 2017 Aug;215:55-61. doi: 10.1016/j.ejogrb.2017.06.005. Epub 2017 Jun 4. PMID 28601728
- [Background] Ovarian Tumor Tissue Analysis (OTTA) Consortium; Goode EL, Block MS, Kalli KR, Vierkant RA, Chen W, Fogarty ZC, Gentry-Maharaj A, Toloczko A, Hein A, Bouligny AL, Jensen A, Osorio A, Hartkopf A, Ryan A, Chudecka-Glaz A, Magliocco AM, Hartmann A, Jung AY, Gao B, Hernandez BY, Fridley BL, McCauley BM, Kennedy CJ, Wang C, Karpinskyj C, de Sousa CB, Tiezzi DG, Wachter DL, Herpel E, Taran FA, Modugno F, Nelson G, Lubinski J, Menkiszak J, Alsop J, Lester J, Garcia-Donas J, Nation J, Hung J, Palacios J, Rothstein JH, Kelley JL, de Andrade JM, Robles-Diaz L, Intermaggio MP, Widschwendter M, Beckmann MW, Ruebner M, Jimenez-Linan M, Singh N, Oszurek O, Harnett PR, Rambau PF, Sinn P, Wagner P, Ghatage P, Sharma R, Edwards RP, Ness RB, Orsulic S, Brucker SY, Johnatty SE, Longacre TA, Ursula E, McGuire V, Sieh W, Natanzon Y, Li Z, Whittemore AS, Anna A, Staebler A, Karlan BY, Gilks B, Bowtell DD, Hogdall E, Candido dos Reis FJ, Steed H, Campbell IG, Gronwald J, Benitez J, Koziak JM, Chang-Claude J, Moysich KB, Kelemen LE, Cook LS, Goodman MT, Garcia MJ, Fasching PA, Kommoss S, Deen S, Kjaer SK, Menon U, Brenton JD, Pharoah PDP, Chenevix-Trench G, Huntsman DG, Winham SJ, Kobel M, Ramus SJ. Dose-Response Association of CD8+ Tumor-Infiltrating Lymphocytes and Survival Time in High-Grade Serous Ovarian Cancer. JAMA Oncol. 2017 Dec 1;3(12):e173290. doi: 10.1001/jamaoncol.2017.3290. PMID 29049607
- [Background] Dai D, Liu L, Huang H, Chen S, Chen B, Cao J, Luo X, Wang F, Luo R, Liu J. Nomograms to Predict the Density of Tumor-Infiltrating Lymphocytes in Patients With High-Grade Serous Ovarian Cancer. Front Oncol. 2021 Feb 25;11:590414. doi: 10.3389/fonc.2021.590414. eCollection 2021. PMID 33718143
- [Background] Lou E, Vogel RI, Hoostal S, Klein M, Linden MA, Teoh D, Geller MA. Tumor-Stroma Proportion as a Predictive Biomarker of Resistance to Platinum-Based Chemotherapy in Patients With Ovarian Cancer. JAMA Oncol. 2019 Aug 1;5(8):1222-1224. doi: 10.1001/jamaoncol.2019.1943. PMID 31152668
- [Background] Qayyum A, Coakley FV, Westphalen AC, Hricak H, Okuno WT, Powell B. Role of CT and MR imaging in predicting optimal cytoreduction of newly diagnosed primary epithelial ovarian cancer. Gynecol Oncol. 2005 Feb;96(2):301-6. doi: 10.1016/j.ygyno.2004.06.054. PMID 15661212
- [Background] Pannu HK, Bristow RE, Montz FJ, Fishman EK. Multidetector CT of peritoneal carcinomatosis from ovarian cancer. Radiographics. 2003 May-Jun;23(3):687-701. doi: 10.1148/rg.233025105. PMID 12740470
- [Background] Avesani G, Arshad M, Lu H, Fotopoulou C, Cannone F, Melotti R, Aboagye E, Rockall A. Radiological assessment of Peritoneal Cancer Index on preoperative CT in ovarian cancer is related to surgical outcome and survival. Radiol Med. 2020 Aug;125(8):770-776. doi: 10.1007/s11547-020-01170-6. Epub 2020 Apr 1. PMID 32239470
- [Background] Engbersen MP, Van' T Sant I, Lok C, Lambregts DMJ, Sonke GS, Beets-Tan RGH, van Driel WJ, Lahaye MJ. MRI with diffusion-weighted imaging to predict feasibility of complete cytoreduction with the peritoneal cancer index (PCI) in advanced stage ovarian cancer patients. Eur J Radiol. 2019 May;114:146-151. doi: 10.1016/j.ejrad.2019.03.007. Epub 2019 Mar 15. PMID 31005166
- [Background] Tardieu M, Lakhman Y, Khellaf L, Cardoso M, Sgarbura O, Colombo PE, Crispin-Ortuzar M, Sala E, Goze-Bac C, Nougaret S. Assessing Histology Structures by Ex Vivo MR Microscopy and Exploring the Link Between MRM-Derived Radiomic Features and Histopathology in Ovarian Cancer. Front Oncol. 2022 Jan 19;11:771848. doi: 10.3389/fonc.2021.771848. eCollection 2021. PMID 35127479
- [Background] Michielsen K, Vergote I, Op de Beeck K, Amant F, Leunen K, Moerman P, Deroose C, Souverijns G, Dymarkowski S, De Keyzer F, Vandecaveye V. Whole-body MRI with diffusion-weighted sequence for staging of patients with suspected ovarian cancer: a clinical feasibility study in comparison to CT and FDG-PET/CT. Eur Radiol. 2014 Apr;24(4):889-901. doi: 10.1007/s00330-013-3083-8. Epub 2013 Dec 11. PMID 24322510
- [Background] Zwanenburg A, Vallieres M, Abdalah MA, Aerts HJWL, Andrearczyk V, Apte A, Ashrafinia S, Bakas S, Beukinga RJ, Boellaard R, Bogowicz M, Boldrini L, Buvat I, Cook GJR, Davatzikos C, Depeursinge A, Desseroit MC, Dinapoli N, Dinh CV, Echegaray S, El Naqa I, Fedorov AY, Gatta R, Gillies RJ, Goh V, Gotz M, Guckenberger M, Ha SM, Hatt M, Isensee F, Lambin P, Leger S, Leijenaar RTH, Lenkowicz J, Lippert F, Losnegard A, Maier-Hein KH, Morin O, Muller H, Napel S, Nioche C, Orlhac F, Pati S, Pfaehler EAG, Rahmim A, Rao AUK, Scherer J, Siddique MM, Sijtsema NM, Socarras Fernandez J, Spezi E, Steenbakkers RJHM, Tanadini-Lang S, Thorwarth D, Troost EGC, Upadhaya T, Valentini V, van Dijk LV, van Griethuysen J, van Velden FHP, Whybra P, Richter C, Lock S. The Image Biomarker Standardization Initiative: Standardized Quantitative Radiomics for High-Throughput Image-based Phenotyping. Radiology. 2020 May;295(2):328-338. doi: 10.1148/radiol.2020191145. Epub 2020 Mar 10. PMID 32154773
- [Background] Lambin P, Leijenaar RTH, Deist TM, Peerlings J, de Jong EEC, van Timmeren J, Sanduleanu S, Larue RTHM, Even AJG, Jochems A, van Wijk Y, Woodruff H, van Soest J, Lustberg T, Roelofs E, van Elmpt W, Dekker A, Mottaghy FM, Wildberger JE, Walsh S. Radiomics: the bridge between medical imaging and personalized medicine. Nat Rev Clin Oncol. 2017 Dec;14(12):749-762. doi: 10.1038/nrclinonc.2017.141. Epub 2017 Oct 4. PMID 28975929
- [Background] van Griethuysen JJM, Fedorov A, Parmar C, Hosny A, Aucoin N, Narayan V, Beets-Tan RGH, Fillion-Robin JC, Pieper S, Aerts HJWL. Computational Radiomics System to Decode the Radiographic Phenotype. Cancer Res. 2017 Nov 1;77(21):e104-e107. doi: 10.1158/0008-5472.CAN-17-0339. PMID 29092951
- [Background] Himoto Y, Veeraraghavan H, Zheng J, Zamarin D, Snyder A, Capanu M, Nougaret S, Vargas HA, Shitano F, Callahan M, Wang W, Sala E, Lakhman Y. Computed Tomography-Derived Radiomic Metrics Can Identify Responders to Immunotherapy in Ovarian Cancer. JCO Precis Oncol. 2019 Aug 15;3:PO.19.00038. doi: 10.1200/PO.19.00038. eCollection 2019. PMID 32914033
- [Background] Bankhead P, Loughrey MB, Fernandez JA, Dombrowski Y, McArt DG, Dunne PD, McQuaid S, Gray RT, Murray LJ, Coleman HG, James JA, Salto-Tellez M, Hamilton PW. QuPath: Open source software for digital pathology image analysis. Sci Rep. 2017 Dec 4;7(1):16878. doi: 10.1038/s41598-017-17204-5. PMID 29203879
- [Background] Simidjievski N, Bodnar C, Tariq I, Scherer P, Andres Terre H, Shams Z, Jamnik M, Lio P. Variational Autoencoders for Cancer Data Integration: Design Principles and Computational Practice. Front Genet. 2019 Dec 11;10:1205. doi: 10.3389/fgene.2019.01205. eCollection 2019. PMID 31921281
- [Background] Weigelt B, Vargas HA, Selenica P, Geyer FC, Mazaheri Y, Blecua P, Conlon N, Hoang LN, Jungbluth AA, Snyder A, Ng CKY, Papanastasiou AD, Sosa RE, Soslow RA, Chi DS, Gardner GJ, Shen R, Reis-Filho JS, Sala E. Radiogenomics Analysis of Intratumor Heterogeneity in a Patient With High-Grade Serous Ovarian Cancer. JCO Precis Oncol. 2019 Jun 6;3:PO.18.00410. doi: 10.1200/PO.18.00410. eCollection 2019. No abstract available. PMID 32914032